CLINICAL TRIAL: NCT05004961
Title: The Performance of Multi-tracer Multimodality PET in Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xuejuan Wang, Principal Investigator, Peking University Cancer Hospital & Institute
Other Study IDs: XW-MMPET-001
Record Dates: First submitted 2021-08-07; First posted 2021-08-13 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Positron-Emission Tomography
Keywords: Positron-Emission Tomography; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigating the performance of Multi-tracer Multimodality PET in lymphoma

DETAILED DESCRIPTION:
In this study investigators evaluated Nodal and Extranodal Lymphoma Lesions uptake by different molecular probe such as FDG, FAPI-04 via multimodality PET (PET/CT and PET/MR). Our Previous studies have shown that uptake of FAPI-04 on PET may be an indicator of lymphoma lesions. The combination of PET with CT/MR allows for depicting metabolic, functional and morphological properties of tumor lesions at the same time, which is therefore an alternative attractive pairing for diagnosis, staging and prognosis of lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed as lymphoma;
* Written informed consent for receiving FAPI-04 PET examinations.
* cancer planned chemotherapy or immunotherapy scheme.
* expected survival ≥ 12 weeks

Exclusion Criteria:

* cannot lie supine for half an hour;
* refuse to join the clinical researcher;
* severe liver or kidney dysfunction
* pregnancy or lactation

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients pathologically diagnosed as lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax | 150 days
  Standardized uptake value of 68Ga/ 18F-NOTA-FAPI 04 for target lesion of subject or suspected tumor in each time point window (SUV)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Zhi, PhD, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Yuan T, Wei M, Yu B, Zhou N, Zhu H, Yang Z, Wang X. Diagnostic performance of integrated whole-body 18F-FDG PET/MRI for detecting bone marrow involvement in indolent lymphoma: Comparison with 18F-FDG PET or MRI alone. Front Oncol. 2023 Mar 13;13:1136687. doi: 10.3389/fonc.2023.1136687. eCollection 2023. PMID 36994205